CLINICAL TRIAL: NCT01033825
Title: A 6-Week Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Safety and Efficacy Study of the Potential Inhibitory Effects on the Hypothalamic-Pituitary-Adrenal Axis of Ciclesonide HFA Nasal Aerosol and Ciclesonide Aqueous Nasal Spray in Subjects 12 Years and Older With Perennial Allergic Rhinitis
Brief Title: Study of the Effects of Ciclesonide Hydrofluoroalkane (HFA) Nasal Aerosol on Hypothalamic-Pituitary-Adrenal (HPA) Axis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060-610
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2012-07-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — ciclesonide; Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Ciclesonide HFA Nasal Aerosol 320 mcg (Experimental): Ciclesonide HFA Nasal Aerosol 320 mcg once daily
  Interventions: Drug: Ciclesonide HFA Nasal Aerosol 320 mcg
- Ciclesonide HFA Nasal Aerosol 160 mcg (Experimental): Ciclesonide HFA Nasal Aerosol 160 mcg once daily
  Interventions: Drug: Ciclesonide HFA Nasal Aerosol 160 mcg
- HFA Nasal Aerosol placebo (Placebo Comparator): HFA Nasal Aerosol Placebo once daily
  Interventions: Drug: HFA Nasal Aerosol placebo
- Ciclesonide Aqueous Nasal Spray 200 mcg (Experimental): Ciclesonide Aqueous Nasal Spray 200 mcg once daily
  Interventions: Drug: Ciclesonide Aqueous Nasal Spray 200 mcg
- AQ Nasal Spray Placebo (Placebo Comparator): AQ Nasal Spray Placebo once daily
  Interventions: Drug: AQ Nasal Spray Placebo
- Placebo HFA plus Dexamethasone 6 mcg (Active Comparator): Placebo HFA plus Dexamethasone 6 mg once daily
  Interventions: Drug: Placebo plus Dexamethasone HFA
- Placebo AQ plus Dexamethasone 6 mg (Active Comparator): Placebo AQ plus Dexamethasone 6 mg once daily
  Interventions: Drug: Placebo AQ plus Dexamethasone 6 mg

INTERVENTIONS:
Drug: Ciclesonide HFA Nasal Aerosol 320 mcg — Ciclesonide HFA Nasal Aerosol 320 μg once daily
  Arms: Ciclesonide HFA Nasal Aerosol 320 mcg
Drug: Ciclesonide HFA Nasal Aerosol 160 mcg — Ciclesonide HFA Nasal Aerosol 160 μg once daily
  Arms: Ciclesonide HFA Nasal Aerosol 160 mcg
Drug: HFA Nasal Aerosol placebo — HFA Nasal Aerosol placebo once daily
  Arms: HFA Nasal Aerosol placebo
Drug: Ciclesonide Aqueous Nasal Spray 200 mcg — Ciclesonide Aqueous Nasal Spray 200 mcg once daily
  Other Names: Omnaris
  Arms: Ciclesonide Aqueous Nasal Spray 200 mcg
Drug: AQ Nasal Spray Placebo — AQ Nasal Spray Placebo once daily
  Arms: AQ Nasal Spray Placebo
Drug: Placebo plus Dexamethasone HFA — Dexamethasone capsules 6 mg once daily
  Other Names: Decadron
  Arms: Placebo HFA plus Dexamethasone 6 mcg
Drug: Placebo AQ plus Dexamethasone 6 mg — Placebo AQ plus Dexamethasone 6 mcg capsules once daily
  Arms: Placebo AQ plus Dexamethasone 6 mg

SUMMARY:
To demonstrate the effects of ciclesonide applied as a nasal aerosol and ciclesonide aqueous (AQ) nasal spray on hypothalamic-pituitary-adrenal axis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, safety and efficacy study of the effects of ciclesonide HFA nasal aerosol and ciclesonide AQ nasal spray on the HPA axis, when administered once daily to male and female subjects 12 years or older diagnosed with Perennial Allergic Rhinitis (PAR). The study consists of a screening period, a single blind run in period, a 6 week double blind treatment period including an active control segment, and a follow up period.

Placebo was used as the control during the double-blind treatment period for both delivery methods (HFA nasal aerosol and aqueous nasal spray)and for the study outcome analyses. There was also a positive control administered to a subset of these placebo subjects during the last 4 days of Week 6 (dexamethasone placebo or dexamethasone 6 mg). The active control was utilized to validate the assay sensitivity (ie, distinguish an effective from an ineffective drug) of this study, as dexamethasone is a known HPA axis suppressant, therefore this subset of placebo subjects was not included in the study outcome analyses.

This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent and assent, including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the Investigator) based on screening physical examination, medical history, and clinical laboratory values (Hematology, Chemistries and Urinalysis).
* If any of the screening Hematology, Chemistries, or Urinalysis are not within the clinical laboratory's reference range, then the subject can be included only if the Investigator judges the deviations to be not clinically significant.
* A history of PAR to a relevant perennial allergen (house dust mites, cockroach, molds, animal dander) for a minimum of two years immediately preceding the study Screening visit. The PAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past and require treatment throughout the entire study period.
* A demonstrated sensitivity to at least one allergen known to induce PAR (house dust mite, animal dander, cockroach, and molds) based on a documented result with a standard skin-prick test either within 90 days prior to screening or performed at the Screening visit. A positive test is defined as a wheal diameter at least 3 mm larger than the negative control wheal for the skin prick test. The subject's positive allergen test must be consistent with the medical history of PAR and must be present in the subject's environment throughout the study.
* Subject, if female, must have a negative serum pregnancy test at screening. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control.

  1. An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following study participation.
  2. Barrier method of contraception, eg, condom and/or diaphragm with spermicide while participating in the study.
  3. Abstinence.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations; recent nasal biopsy; nasal trauma; or nasal ulcers or perforations. Surgery and atrophic rhinitis or rhinitis medicamentosa are not permitted within the last 120 days prior to the Screening visit.
* Subject is, in the investigator's judgement, having a seasonal exacerbation at the time of screening.
* Participation in any investigational drug trial within the 30 days preceding the Screening visit or planned participation in another investigational drug trial at any time during this trial.
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulation of ciclesonide.
* History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, influenza, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening visit.
* History of alcohol or drug abuse within 2 years preceding the Screening visit.
* History of a positive test for HIV, hepatitis B or hepatitis C.
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta agonists and any controller drugs (eg, theophylline, leukotriene antagonists, etc.); intermittent use (less than or equal to 3 uses per week) of inhaled short acting beta-agonists is acceptable. Use of short acting beta-agonists for exercise-induced bronchospasm will be allowed.
* Expected use of any disallowed concomitant medications during the treatment period.
* Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit and use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
* Previous randomization in an intranasal ciclesonide HFA nasal aerosol study.
* Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit.
* Initiation of pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or planned dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to screening and use of a stable (maintenance) dose during the study period may be considered for inclusion.
* Study participation by clinical investigator site employees and/or their immediate relatives who reside in the same household.
* Study participation by more than one subject from the same household.
* Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial: impaired hepatic function including alcohol related liver disease or cirrhosis; history of ocular disturbances, eg, glaucoma or posterior subcapsular cataracts; any systemic infection hematological, hepatic, renal, endocrine (except for controlled diabetes mellitus or postmenopausal symptoms or hypothyroidism; gastrointestinal disease; malignancy (excluding basal cell carcinoma); current neuropsychological condition with or without drug therapy
* Any condition that, in the judgment of the investigator, would preclude the subject from completing the protocol with capture of the assessments as written.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneappolis, Minnesota
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo HFA Plus Dexamethasone 6 mg: Placebo HFA plus Dexamethasone 6 mg once daily. Placebo is the study control & used for the study outcome analyses (CIC placebo/DEX placebo) for each delivery method (HFA or AQ). The positive control was used in a subset of the placebo subjects (18 subjects) during the last 4 days of Week 6. The active control was utilized to validate the assay sensitivity of the study, therefore this subset of placebo subjects was not included in the study outcome analyses.
- Placebo AQ Plus Dexamethasone 6 mg: Placebo AQ plus Dexamethasone 6 mg once daily. Placebo is the study control & used for the study outcome analyses (CIC placebo/DEX placebo) for each delivery method (HFA or AQ). The positive control was used in a subset of these placebo subjects (18 subjects) during the last 4 days of Week 6. The active control was utilized to validate the assay sensitivity of the study, therefore this subset of placebo subjects was not included in the study outcome analyses.
Period: Overall Study
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo | Placebo HFA Plus Dexamethasone 6 mg | Placebo AQ Plus Dexamethasone 6 mg
Started | 51 | 60 | 57 | 48 | 58 | 18 | 18
Completed | 48 | 57 | 55 | 46 | 56 | 18 | 18
Not Completed | 3 | 3 | 2 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo | Placebo HFA Plus Dexamethasone 6 mg | Placebo AQ Plus Dexamethasone 6 mg | Total
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58 | 18 | 18 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 10 | 12 | 8 | 9 | 2 | 3 | 48
  Between 18 and 65 years | 47 | 50 | 43 | 40 | 48 | 16 | 15 | 259
  >=65 years | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 35.8 (13.62) | 34.5 (13.42) | 33.0 (15.69) | 32.3 (12.53) | 35.5 (14.55) | 35.4 (12.94) | 34.0 (134.41) | 34.26 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 37 | 30 | 33 | 6 | 12 | 187
  Male | 19 | 23 | 20 | 18 | 25 | 12 | 6 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 16 | 6 | 11 | 10 | 3 | 3 | 60
  Not Hispanic or Latino | 40 | 44 | 51 | 37 | 48 | 15 | 15 | 250
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, customized [Number; unit: particpants]
  White/Caucasian | 49 | 51 | 52 | 42 | 52 | 15 | 15 | 276
  Black or African American | 1 | 4 | 5 | 4 | 5 | 2 | 1 | 22
  Asian | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 6
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Multiple | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Serum Cortisol Area Under the Concentration-time Curve (AUC)(0-24h) at Baseline
Description: AUC(0-24h) will be computed using the linear trapezoidal rule based on the actual time of serum cortisol drawing. AUC(0-24) is then approximated by the sum of the areas of trapezoids. The trapezoid for each time interval is based on the actual times of non-missing cortisol values, and is defined by the actual time interval as the base, the line connecting the two cortisol values, and the two vertical sides at the two time points. Raw data is presented for baseline values (i.e. mean/SD), while inferential statistics are presented for week 6 values (i.e. LS mean/SE).
Time Frame: Baseline
Population: Per Protocol Population. Analysis does not include the subjects that received Dexamethasone during the active control period.
Measure: Mean (Standard Deviation); unit: mcg•h/dL
Groups:
- Ciclesonide HFA Nasal Aerosol 320 Mcg: Ciclesonide hydrofluoroalkane (HFA) Nasal Aerosol 320 mcg once daily
- Ciclesonide Aqueous Nasal Spray 200 Mcg: Ciclesonide Aqueous (AQ) Nasal Spray 200 mcg once daily
- Placebo Aqueous Nasal Spray: AQ Nasal Spray Placebo once daily
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | Placebo Aqueous Nasal Spray
Number analyzed (Participants) | 50 | 60 | 57 | 48 | 58
mcg•h/dL | 183.2 (61.9) | 171.7 (40.1) | 173.1 (53.5) | 172.8 (42.5) | 179.0 (37.9)

2. Secondary Outcome: Number of Subjects Experiencing Adverse Events (AEs)
Time Frame: Weeks 0-6
Population: Intent to Treat Population.
Measure: Number; unit: participants
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | Placebo Aqueous Nasal Spray
Number analyzed (Participants) | 51 | 60 | 75 | 48 | 76
participants | 23 | 17 | 23 | 19 | 29

3. Secondary Outcome: Percentage of Subjects Experiencing Adverse Events (AEs)
Time Frame: Weeks 0-6
Population: Intent to Treat Population.
Measure: Number; unit: percentage of subjects
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 75 | 48 | 76
percentage of subjects | 45.1 | 28.3 | 30.7 | 39.6 | 38.2

4. Secondary Outcome: Number of Subjects Experiencing Serious Adverse Events (SAEs).
Time Frame: Weeks 0-6
Population: Intent to Treat Population.
Measure: Number; unit: participants
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 48 | 57 | 75 | 47 | 76
participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Subjects Experiencing Serious Adverse Events (SAEs).
Time Frame: Weeks 0-6
Population: Intent to Treat Population
Measure: Number; unit: percentage of subjects
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 48 | 57 | 75 | 47 | 76
percentage of subjects | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Subjects Who Discontinue Due to AEs
Time Frame: Weeks 0-6
Population: Intent to Treat Population.
Measure: Number; unit: participants
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 75 | 48 | 76
participants | 0 | 0 | 0 | 1 | 0

7. Secondary Outcome: Percentage of Subjects Who Discontinue Due to AEs
Time Frame: Weeks 0-6
Population: Intent to Treat Population
Measure: Number; unit: percentage of subjects
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 48 | 57 | 75 | 47 | 76
percentage of subjects | 0 | 0 | 0 | 2.1 | 0

8. Secondary Outcome: Number of Subjects Experiencing Local Nasal AEs
Description: Local Nasal adverse events are defined as adverse events occurring in the middle ear, nose, throat, and upper respiratory tract down to the larynx, anatomic regions.
Time Frame: Weeks 0-6
Population: Intent to Treat Population
Measure: Number; unit: participants
Groups:
- Placebo HFA Plus 6 mg Dexamethasone: Placebo HFA plus 6 mg Dexamethasone once daily
- Placebo AQ Plus 6 mg Dexamethasone: Placebo AQ plus 6 mg Dexamethasone once daily
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo | Placebo HFA Plus 6 mg Dexamethasone | Placebo AQ Plus 6 mg Dexamethasone
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58 | 18 | 18
participants | 21 | 11 | 8 | 16 | 11 | 5 | 1

9. Secondary Outcome: Percentage of Subjects Experiencing Local Nasal AEs
Description: as for outcome 8
Time Frame: Weeks 0-6
Population: Intent to Treat Population
Measure: Number; unit: percentage of subjects
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo | Placebo HFA Plus 6 mg Dexamethasone | Placebo AQ Plus 6 mg Dexamethasone
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58 | 18 | 18
percentage of subjects | 41.2 | 18.3 | 14.0 | 33.3 | 19.0 | 27.8 | 5.6

10. Secondary Outcome: Serum Cortisol Area Under the Concentration-time Curve (AUC)(0-12h) at Baseline
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg•h/dL
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
mcg•h/dL | 99.8 (38.3) | 95.1 (28.5) | 92.0 (31.3) | 91.9 (25.8) | 97.2 (25.0)

11. Secondary Outcome: Change in Serum Cortisol Area Under the Concentration-time Curve (AUC)(0-12h) From Baseline After 6 Weeks of Treatment
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mcg•h/dL
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
mcg•h/dL | -1.0 (3.2) | -1.3 (3.0) | 0.5 (3.0) | -5.8 (3.0) | -2.9 (2.7)

12. Secondary Outcome: Serum Cortisol Area Under the Concentration-time Curve (AUC)(12-24h) at Baseline
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg•h/dL
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
mcg•h/dL | 83.4 (30.2) | 76.2 (24.0) | 81.1 (28.7) | 80.9 (26.8) | 81.8 (22.8)

13. Secondary Outcome: Change in Serum Cortisol Area Under the Concentration-time Curve (AUC)(12-24h) From Baseline After 6 Weeks of Treatment
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mcg•h/dL
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
mcg•h/dL | -3.9 (2.9) | -2.0 (2.7) | -5.9 (2.7) | -6.1 (3.7) | 2.2 (3.4)

14. Secondary Outcome: Baseline Daily Subject-reported AM Reflective TNSS
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale | 7.55 (2.39) | 8.03 (2.27) | 7.81 (2.47) | 7.91 (2.50) | 7.84 (2.58)

15. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Reflective TNSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 14
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale | -1.80 (0.29) | -1.75 (0.26) | -0.35 (0.27) | -1.18 (0.30) | -0.91 (0.28)

16. Secondary Outcome: Baseline Daily Subject-reported PM Reflective TNSS
Description: as for outcome 14
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale | 7.82 (2.40) | 8.39 (2.11) | 7.83 (2.52) | 8.13 (2.66) | 8.16 (2.51)

17. Secondary Outcome: Change From Baseline in Daily Subject-reported PM Reflective TNSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 14
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale | -1.77 (0.30) | -1.88 (0.28) | -0.31 (0.28) | -1.14 (0.29) | -1.19 (0.26)

18. Secondary Outcome: Baseline Daily Subject-reported AM Instantaneous TNSS
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptom on a scale of 0-3 where:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale | 6.91 (2.68) | 7.63 (2.35) | 7.37 (2.68) | 7.24 (2.43) | 7.19 (2.84)

19. Secondary Outcome: Change From Baseline in Daily Subject-reported AM Instantaneous TNSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 18
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale | -1.52 (0.27) | -1.62 (0.25) | -0.26 (0.25) | -1.23 (0.29) | -0.60 (0.26)

20. Secondary Outcome: Baseline Daily Subject-reported AM and PM Reflective TNSS
Description: as for outcome 14
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
units on a scale | 7.68 (2.33) | 8.20 (2.14) | 7.82 (2.45) | 8.01 (2.52) | 8.01 (2.49)

21. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM Reflective TNSS Averaged Over Each Week, and Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 14
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
units on a scale | -1.78 (0.29) | -1.82 (0.27) | -0.33 (0.27) | -1.16 (0.29) | -1.06 (0.27)

22. Secondary Outcome: Baseline Daily Subject-reported PM Instantaneous TNSS
Description: as for outcome 18
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale | 6.84 (3.09) | 7.60 (2.37) | 7.13 (2.75) | 7.38 (2.68) | 7.44 (2.74)

23. Secondary Outcome: Change From Baseline in Daily Subject-reported PM Instantaneous TNSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 18
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale | -1.39 (0.28) | -1.67 (0.26) | -0.10 (0.26) | -1.09 (0.30) | -0.88 (0.28)

24. Secondary Outcome: Baseline Daily Subject-reported AM and PM Instantaneous TNSS
Description: as for outcome 18
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
units on a scale | 6.87 (2.84) | 7.62 (2.29) | 7.26 (2.67) | 7.30 (2.52) | 7.33 (2.74)

25. Secondary Outcome: Change From Baseline in Daily Subject-reported AM and PM Instantaneous TNSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 18
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
units on a scale | -1.45 (0.27) | -1.67 (0.25) | -0.19 (0.25) | -1.15 (0.29) | -0.75 (0.27)

26. Secondary Outcome: Baseline Daily Subject-reported Individual AM Reflective NSS
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent (no sign/symptom evident);
  1. = mild
  2. = moderate
  3. = severe Reflective NSS measures these symptoms over the previous 12-hour time interval. Difference was calculated by subtracting baseline value from the 6-week DB average. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale
  Baseline Nasal Sneezing | 1.56 (0.83) | 1.65 (0.88) | 1.54 (0.89) | 1.42 (0.81) | 1.57 (0.93)
  Baseline Runny Nose | 1.99 (0.68) | 2.16 (0.63) | 2.15 (0.70) | 2.27 (0.71) | 2.06 (0.76)
  Baseline Nasal Itching | 1.71 (0.85) | 1.89 (0.75) | 1.83 (0.83) | 1.85 (0.85) | 1.92 (0.83)
  Baseline Nasal Congestion | 2.30 (0.59) | 2.32 (0.57) | 2.29 (0.60) | 2.36 (0.66) | 2.29 (0.62)

27. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM Reflective NSS Averaged Over the 6 Weeks of Double-blind Treatment Period
Description: as for outcome 26
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale
  Nasal Sneezing | -0.41 (0.09) | -0.41 (0.08) | -0.09 (0.08) | -0.28 (0.08) | -0.25 (0.08)
  Runny Nose | -0.50 (0.08) | -0.50 (0.08) | -0.17 (0.08) | -0.36 (0.10) | -0.29 (0.09)
  Nasal Itching | -0.40 (0.08) | -0.40 (0.08) | -0.05 (0.08) | -0.33 (0.09) | -0.25 (0.08)
  Nasal Congestion | -0.49 (0.07) | -0.42 (0.07) | -0.05 (0.07) | -0.20 (0.09) | -0.13 (0.08)

28. Secondary Outcome: Baseline Daily Subject-reported Individual PM Reflective NSS
Description: as for outcome 26
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale
  Baseline Nasal Sneezing | 1.82 (0.71) | 1.87 (0.76) | 1.69 (0.81) | 1.59 (0.83) | 1.74 (0.87)
  Baseline Runny Nose | 2.03 (0.66) | 2.20 (0.58) | 2.11 (0.71) | 2.30 (0.74) | 2.16 (0.73)
  Baseline Nasal Itching | 1.75 (0.83) | 2.02 (0.75) | 1.80 (0.82) | 1.93 (0.87) | 2.00 (0.78)
  Baseline Nasal Congestion | 2.23 (0.72) | 2.30 (0.54) | 2.23 (0.67) | 2.31 (0.73) | 2.25 (0.63)

29. Primary Outcome: The Change in Serum Cortisol Area Under the Concentration-time Curve (AUC)(0-24h) From Baseline to Week 6 of the Double Blind Treatment Period
Description: Change is calculated as week 6 minus baseline. AUC(0-24h) will be computed using the linear trapezoidal rule based on the actual time of serum cortisol drawing. AUC(0-24) is then approximated by the sum of the areas of trapezoids. The trapezoid for each time interval is based on the actual times of non-missing cortisol values, and is defined by the actual time interval as the base, the line connecting the two cortisol values, and the two vertical sides at the two time points. Raw data is presented for baseline values (i.e. mean/SD), while inferential statistics are presented for week 6 values (i.e. LS mean/SE).
Time Frame: week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mcg•h/dL
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | Placebo Aqueous Nasal Spray
Number analyzed (Participants) | 50 | 60 | 57 | 48 | 58
mcg•h/dL | -4.6 (5.0) | -2.6 (4.6) | -5.0 (4.6) | -11.4 (5.7) | -1.0 (5.2)
Statistical Analysis 1: Comparison: Ciclesonide HFA Nasal Aerosol 320 Mcg vs HFA Nasal Aerosol Placebo; Standard bioequivalence bounds of a 20% difference based on the clinical judgment was used to determine the delta; Test type: Non-Inferiority or Equivalence — Non-inferiority will be demonstrated if the 95% CI upper bound for the difference between ciclesonide and placebo with placebo dexamethasone (placebo minus ciclesonide) is <Margin. In order to have 90% power to demonstrate non-inferiority of ciclesonide 320 μg to HFA placebo, 46 evaluable subjects per group are needed using a 1-sided alpha level of 0.025, a standard deviation of 55 μg h/dL, a non-inferiority margin of 38 μh /dL, assuming no true difference exists; p > 0.05, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-13.9 to 13.0] — Null Hypothesis: the difference in serum cortisol levels between placebo and active (placebo-active)>=38 Alternative Hypothesis: the difference in serum cortisol levels between placebo and active (placebo-active)<38
Statistical Analysis 2: Comparison: Ciclesonide HFA Nasal Aerosol 160 Mcg vs HFA Nasal Aerosol Placebo; Standard bioequivalence bounds of a 20% difference based on the clinical judgment was used to determine the delta; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 29, analysis 1]; p = 0.025, ANCOVA; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-15.1 to 10.2]
Statistical Analysis 3: Comparison: Ciclesonide Aqueous Nasal Spray 200 Mcg vs Placebo Aqueous Nasal Spray; Standard bioequivalence bounds of a 20% difference based on the clinical judgment was used to determine the delta; Test type: Non-Inferiority or Equivalence — Non-inferiority will be demonstrated if the 95% CI upper bound for the difference between ciclesonide and placebo with placebo dexamethasone (placebo minus ciclesonide) is <Margin. In order to have 90% power to demonstrate non-inferiority of ciclesonide nasal spray 200 μg to placebo nasal spray 46 evaluable (per protocol) subjects per group are needed using a 1-sided alpha level of 0.025, a standard deviation of 55 μg h/dL, a non-inferiority margin of 38 μh /dL; p > 0.05, ANCOVA; Mean Difference (Final Values) = 10.4, 95% CI 2-sided [-4.7 to 25.5]

30. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual PM Reflective NSS Averaged Over the 6 Weeks of Double-blind Treatment Period
Description: as for outcome 26
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale
  Nasal Sneezing | -0.45 (0.09) | -0.48 (0.08) | -0.13 (0.08) | -0.23 (0.08) | -0.27 (0.08)
  Runny Nose | -0.49 (0.08) | -0.48 (0.08) | -0.09 (0.08) | -0.37 (0.09) | -0.37 (0.08)
  Nasal Itching | -0.38 (0.08) | -0.46 (0.08) | -0.05 (0.08) | -0.32 (0.09) | -0.34 (0.08)
  Nasal Congestion | -0.44 (0.08) | -0.44 (0.07) | -0.04 (0.07) | -0.20 (0.09) | -0.21 (0.08)

31. Secondary Outcome: Baseline Daily Subject-reported Individual AM and PM Reflective NSS
Description: as for outcome 26
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
units on a scale
  Baseline Nasal Sneezing | 1.69 (0.73) | 1.76 (0.79) | 1.62 (0.83) | 1.51 (0.78) | 1.66 (0.87)
  Baseline Runny Nose | 2.01 (0.65) | 2.18 (0.59) | 2.13 (0.69) | 2.29 (0.70) | 2.11 (0.72)
  Baseline Nasal Itching | 1.73 (0.83) | 1.95 (0.73) | 1.82 (0.80) | 1.89 (0.85) | 1.96 (0.79)
  Baseline Nasal Congestion | 2.26 (0.63) | 2.31 (0.53) | 2.26 (0.62) | 2.33 (0.67) | 2.27 (0.61)

32. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM and PM Reflective NSS Averaged Over the 6 Weeks of Double-blind Treatment Period
Description: as for outcome 26
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
units on a scale
  Nasal Sneezing | -0.43 (0.09) | -0.45 (0.08) | -0.11 (0.08) | -0.25 (0.08) | -0.26 (0.07)
  Runny Nose | -0.50 (0.08) | -0.50 (0.07) | -0.13 (0.08) | -0.37 (0.09) | -0.33 (0.08)
  Nasal Itching | -0.39 (0.08) | -0.43 (0.08) | -0.05 (0.08) | -0.32 (0.09) | -0.30 (0.08)
  Nasal Congestion | -0.47 (0.07) | -0.43 (0.07) | -0.04 (0.07) | -0.20 (0.09) | -0.17 (0.08)

33. Secondary Outcome: Baseline Daily Subject-reported Individual AM Instantaneous NSS
Description: NSS is the assessment of the individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent (no sign/symptom evident);
  1. = mild
  2. = moderate
  3. = severe Instantaneous NSS measures these symptoms over the previous 10 minute time interval. Difference was calculated by subtracting baseline value from the 6-week DB average. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale
  Baseline Nasal Sneezing | 1.24 (0.82) | 1.43 (0.96) | 1.34 (0.94) | 1.15 (0.85) | 1.30 (1.02)
  Baseline Runny Nose | 1.83 (0.84) | 2.08 (0.66) | 2.01 (0.74) | 2.08 (0.68) | 1.93 (0.89)
  Baseline Nasal Itching | 1.61 (0.86) | 1.85 (0.75) | 1.76 (0.89) | 1.76 (0.89) | 1.76 (0.91)
  Baseline Nasal Congestion | 2.24 (0.67) | 2.27 (0.58) | 2.27 (0.60) | 2.25 (0.66) | 2.20 (0.66)

34. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM Instantaneous NSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 33
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale
  Nasal Sneezing | -0.32 (0.08) | -0.37 (0.07) | -0.06 (0.08) | -0.24 (0.08) | -0.17 (0.07)
  Runny Nose | -0.43 (0.08) | -0.47 (0.08) | -0.12 (0.08) | -0.36 (0.10) | -0.23 (0.09)
  Nasal Itching | -0.38 (0.08) | -0.40 (0.07) | -0.03 (0.08) | -0.40 (0.09) | -0.14 (0.08)
  Nasal Congestion | -0.41 (0.07) | -0.37 (0.07) | -0.05 (0.07) | -0.20 (0.08) | -0.06 (0.07)

35. Secondary Outcome: Baseline Daily Subject-reported Individual PM Instantaneous NSS
Description: as for outcome 33
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale
  Baseline Nasal Sneezing | 1.42 (0.89) | 1.51 (0.86) | 1.40 (0.93) | 1.30 (0.85) | 1.47 (0.92)
  Baseline Runny Nose | 1.80 (0.85) | 2.03 (0.73) | 1.98 (0.72) | 2.13 (0.75) | 2.01 (0.76)
  Baseline Nasal Itching | 1.60 (0.90) | 1.88 (0.78) | 1.64 (0.84) | 1.79 (0.87) | 1.84 (0.91)
  Baseline Nasal Congestion | 2.02 (0.82) | 2.19 (0.59) | 2.11 (0.68) | 2.16 (0.76) | 2.12 (0.65)

36. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual PM Instantaneous NSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 33
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 50 | 59 | 57 | 48 | 58
units on a scale
  Nasal Sneezing | -0.33 (0.08) | -0.37 (0.08) | -0.07 (0.08) | -0.24 (0.08) | -0.22 (0.08)
  Runny Nose | -0.41 (0.08) | -0.45 (0.07) | -0.08 (0.08) | -0.33 (0.10) | -0.30 (0.09)
  Nasal Itching | -0.32 (0.08) | -0.44 (0.07) | 0.02 (0.07) | -0.35 (0.09) | -0.25 (0.08)
  Nasal Congestion | -0.34 (0.07) | -0.39 (0.07) | 0.02 (0.07) | -0.15 (0.09) | -0.12 (0.08)

37. Secondary Outcome: Baseline Daily Subject-reported Individual AM and PM Instantaneous NSS
Description: as for outcome 33
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
units on a scale
  Baseline Nasal Sneezing | 1.33 (0.83) | 1.47 (0.89) | 1.37 (0.91) | 1.22 (0.83) | 1.38 (0.95)
  Baseline Runny Nose | 1.81 (0.83) | 2.05 (0.67) | 2.00 (0.72) | 2.10 (0.69) | 1.98 (0.80)
  Baseline Nasal Itching | 1.61 (0.86) | 1.87 (0.75) | 1.70 (0.84) | 1.78 (0.87) | 1.80 (0.89)
  Baseline Nasal Congestion | 2.13 (0.72) | 2.23 (0.55) | 2.19 (0.62) | 2.20 (0.68) | 2.16 (0.63)

38. Secondary Outcome: Change From Baseline in Daily Subject-reported Individual AM and PM Instantaneous NSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: as for outcome 33
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Number analyzed (Participants) | 51 | 60 | 57 | 48 | 58
units on a scale
  Nasal Sneezing | -0.32 (0.08) | -0.37 (0.07) | -0.06 (0.07) | -0.23 (0.08) | -0.20 (0.07)
  Runny Nose | -0.42 (0.08) | -0.47 (0.07) | -0.10 (0.07) | -0.35 (0.09) | -0.27 (0.09)
  Nasal Itching | -0.35 (0.08) | -0.42 (0.07) | -0.01 (0.07) | -0.37 (0.09) | -0.20 (0.08)
  Nasal Congestion | -0.37 (0.07) | -0.39 (0.06) | -0.01 (0.06) | -0.17 (0.08) | -0.09 (0.08)

39. Secondary Outcome: Time to Maximal Effect Over 6 Weeks of Double-blind Treatment.
Description: The time to maximal effect is defined as the number of days until the first treatment day on which the estimated difference between each active treatment group and corresponding placebo is at least 90% of the largest estimated difference. This is based on the analyses of change from baseline in the average of AM and PM reflective TNSS scores for each day. The evaluation is made separately for each dose level of Ciclesonide HFA compared to placebo. Difference is calculated as placebo - ciclesonide. Analysis of HFA data and AQ data were conducted separately.
Time Frame: Weeks 0-6
Population: as for outcome 1
Measure: Number; unit: Number of days
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | Ciclesonide Aqueous Nasal Spray 200 Mcg
Number analyzed (Participants) | 51 | 60 | 48
Number of days | 15 | 29 | 7

40. Secondary Outcome: Ratio (Percentage) of Correct Advances of the Dose Indicator Out of Expected Advances.
Description: Ratio of correct advance is defined as the (number of doses actuated/number of dose reported).
Time Frame: Weeks 1-2, 2-4
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: percentage of correct advances
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo
Number analyzed (Participants) | 51 | 60 | 75
percentage of correct advances
  Weeks 1-2 (n=49,58,75) | 106.3 (10.8) | 106.2 (12.1) | 105.3 (15.8)
  Weeks 2-4 (n=46,52,71) | 105.6 (11.8) | 105.9 (10.5) | 105.8 (11.7)

41. Secondary Outcome: Number of Devices With Actuation Consistency
Description: Actuation consistency is defined as a dose indicator count within ±20% of the subject self report of study medication administration.
Time Frame: Weeks 1-4
Population: Intent to Treat Population
Measure: Number; unit: Devices
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | Ciclesonide Aqueous Nasal Spray 200 Mcg
Number analyzed (Participants) | 46 | 52 | 71
Devices | 42 | 48 | 68

42. Secondary Outcome: Percentage of Devices With Actuation Consistency
Description: as for outcome 41
Time Frame: Weeks 1-4
Population: Intent to Treat Population
Measure: Number; unit: percentage of devices
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo
Number analyzed (Participants) | 46 | 52 | 71
percentage of devices | 91.3 | 92.3 | 95.8

43. Secondary Outcome: Number of Devices With Major Discrepancies
Description: A major discrepancy is defined as a discrepancy of >20 actuations between the dose indicator and subject self report of study medication administration.
Time Frame: Week 6
Population: Intent to Treat Population
Measure: Number; unit: Devices
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | Ciclesonide Aqueous Nasal Spray 200 Mcg
Number analyzed (Participants) | 46 | 52 | 71
Devices | 0 | 2 | 1

44. Secondary Outcome: Percentage of Devices With Major Discrepancies
Description: as for outcome 43
Time Frame: Week 6
Population: Intent to Treat Population
Measure: Number; unit: percentage of devices
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo
Number analyzed (Participants) | 46 | 52 | 71
percentage of devices | 0 | 3.8 | 1.4

ADVERSE EVENTS:
Description: Adverse events were NOT assessed for active control (Placebo plus Dexamethasone) groups.
Arm/Group | Ciclesonide HFA Nasal Aerosol 320 Mcg | Ciclesonide HFA Nasal Aerosol 160 Mcg | HFA Nasal Aerosol Placebo | Ciclesonide Aqueous Nasal Spray 200 Mcg | AQ Nasal Spray Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/57 | 0/18 | 0/47 | 0/57
Other Adverse Events (participants affected / at risk) | 24/51 | 22/60 | 16/57 | 25/48 | 22/58
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide HFA Nasal Aerosol 320 Mcg (N=51) | Ciclesonide HFA Nasal Aerosol 160 Mcg (N=60) | HFA Nasal Aerosol Placebo (N=57) | Ciclesonide Aqueous Nasal Spray 200 Mcg (N=48) | AQ Nasal Spray Placebo (N=58)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyphthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Instillation site discomfort (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myaglia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Drug withdrawal headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 7 (11)
Sinus Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 4 (7) | 3 (3) | 9 (16) | 3 (7)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Dose levels investigated were higher than the US FDA approved dose (74 mcg once daily) for allergic rhinitis subjects. Publication references to 148 and 282mcg are equivalent to 160 and 320mcg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other